CLINICAL TRIAL: NCT06933264
Title: Corporal Composition and Gut Microbiome Modification Through Exclusion Dietary Intervention in Adult Patients With Crohn's Disease: Protocol for a Prospective, Interventional, Controlled, Randomized Clinical Trial
Brief Title: Corporal Composition and Gut Microbiome Modification Through Exclusion Dietary Intervention in Crohn's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Collaborators: Universidad de Murcia (Other); Sociedad Española de Endocrinología y Nutrición (Unknown); Instituto Murciano de Investigación Biosanitaria (IMIB) (Unknown)
Responsible Party: Principal Investigator, Rosario Paloma Cano Mármol, MIR of Endocrinology and Nutrition, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4-10-HCUVA
Record Dates: First submitted 2025-03-23; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
Keywords: Crohn disease; Gut microbiome; Nutrition; Exclusion diet
MeSH Terms: conditions — Crohn Disease | interventions — Elimination Diets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exclusion diet (Experimental): Experimental Group: Patients will receive modifications to their pharmacological and will be assigned to an intervention consisting of an exclusion diet in conjunc-tion with supplemental enteral nutrition. This nutritional strategy will involve a progressive increase in the caloric intake derived from the diet, coupled with a corresponding reduction in supplemental enteral nutrition.
  Interventions: Dietary Supplement: Exclusion diet
- Mediterranean diet (No Intervention): Control Group: Patients will receive modifications to their pharmacological treatment alongside standard nutritional recommendations.

INTERVENTIONS:
Dietary Supplement: Exclusion diet — Experimental Group: Patients will receive modifications to their pharmacological and will be assigned to an intervention consisting of an exclusion diet in conjunc-tion with supplemental enteral nutrition. This nutritional strategy will involve a progressive increase in the caloric intake derived from the diet, coupled with a corresponding reduction in supplemental enteral nutrition.
  Other Names: Experimental group
  Arms: Exclusion diet

SUMMARY:
Crohn's disease (CD) is an inflammatory bowel disease in which there is an alteration of the homeostasis and functionality of the intestinal mucosa accompanied by a dysbiosis of the commensal microbiota. The analysis of different dietary strategies to achieve CD remission and reduce gastrointestinal symptoms concludes that it is nec-essary to restrict the intake of ultra-processed products and to promote the consump-tion of those with anti-inflammatory effects that improve intestinal permeability and dysbiosis. Based on previous studies conducted in other cohorts, mainly paediatric, we propose an experimental, prospective, randomised study in patients with active CD who do not show improvement with conventional pharmacological treatment. The control group will receive standard nutritional recommendations while the interven-tion group will be prescribed an exclusion diet supplemented with enteral nutrition. In the present project we plan to conduct a detailed study to determine the potential of the exclusion diet for the treatment and remission of CD in adult patients, with the hypothesis that this nutritional intervention will be able to modify and improve intes-tinal dysbiosis, inflammatory status and clinical and body composition markers in these patients.

DETAILED DESCRIPTION:
An analysis of various dietary strategies to achieve remission of CD and reduce gastrointestinal symptoms concludes that it is necessary to restrict the intake of ultra-processed products while promoting foods with anti-inflammatory effects that improve intestinal permeability and dysbiosis. The European Society for Clinical Nutrition and Metabolism (ESPEN) acknowledges that there is insufficient evidence to recommend a specific diet and emphasizes the importance of individualization. Current scientific literature supports the use of the exclusion diet (ED) in CD, which is characterized by the exclusion of frozen or packaged foods due to their additive content and the inclusion of fresh, fiber-rich foods-owing to the benefits observed in symptom remission in the pediatric population. However, evidence in adults, although encouraging, remains limited. The ED is supplemented with a specific enteral nutrition formula that should not exceed 1250 Kcal/day and is administered at a proportion of 25-50%, depending on the phase of the diet. The first two phases last 6 weeks each (12 weeks in total) and include foods that must be consumed daily. In the final maintenance phase, starting from week 13, there are no mandatory foods, and a Mediterranean diet is promoted. The literature also advocates for modifying the dietary pattern by reducing ultra-processed foods and adhering to the Mediterranean diet after one year of initiating the ED.

On the other hand, evidence regarding the impact on body composition in patients with CD is scarce and heterogeneous, which justifies further research and the publication of higher-quality data. These findings could present an opportunity to improve the treatment of patients with CD and to incorporate body composition assessment into routine clinical practice.

The primary advantage of this dietary strategy lies in its balanced, sustainable, and palatable nature, making it easier to adhere to over time. This is largely due to its inclusion of dietary fiber and essential substrates necessary for the production of short-chain fatty acids. The exclusion diet is based on the elimination or inclusion of specific dietary components while ensuring a nutrient composition that supports growth and maintenance of lean body mass.

Foods and additives that should be excluded from this diet include those associ-ated with high fat intake (particularly from animal sources, such as red meat), dairy products, wheat, alcohol, yeast, and insoluble fiber. Additionally, food additives recommended for avoidance include emulsifiers, carrageenan, maltodextrins, sulfites, and titanium dioxide. Conversely, the diet should be low in taurine, rich in pro-teins and complex carbohydrates, and free of gluten or modified starches.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes over 18 years of age.
* A diagnosis of active luminal CD with small bowel involvement, with or without colonic involvement, prior to study inclusion.
* Active symptoms of CD at the time of initiation of the nutritional intervention.
* Active disease, defined as a Harvey-Bradshaw Index (HBI) > 4 and an objective measure of disease activity, such as an elevated inflammatory marker (CRP > 5 mg/L or 0.5 mg/dL, or calprotectin ≥ 250 µg/g) and/or a radiological imaging test (MR enterography or intestinal ultrasound) or an endoscopic test (ileocolonoscopy or capsule endoscopy).
* Ability and willingness to adhere to one of the nutritional interventions.
* Capacity to complete and sign the informed consent form.

Exclusion Criteria:

* Patients experiencing a severe flare that is associated with fistulizing tracts or strictures during the study period.
* Hospitalized patients.
* Patients with known intolerance or hypersensitivity to the components of the nu-tritional supplement Modulen IBD.
* Patients following another diet or who are participating in other nutritional trials.
* Patients scheduled for surgical intervention during the study period.
* Patients with active malignancy.
* Patients undergoing treatment with antibiotics or probiotics.
* Patients with other clinical conditions that may interfere with the implementation of the nutritional interventions (such as heart disease, celiac disease, uncontrolled diabetes, active infections, tuberculosis, or a positive stool test for Clostridium dif-ficile toxin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Body composition | From enrollment to the end of study at 24 weeks
  The primary objective of this clinical study is to determine the effectiveness and impact on body composition of implementing an exclusion diet for symptomatic remission in adult patients with active Crohn disease.

SECONDARY OUTCOMES:
Inflamatory parameters | From enrollment to the end of study at 24 weeks
  Inflammatory parameters in blood: C-reactive protein (mg/dl)
Inflamatory parameters | From enrollment to the end of study at 24 weeks
  Inflammatory parameters in blood: Inflammatory parameters in blood: erythrocyte sedimentation rate (mm/h)
Inflamatory parameters | From enrollment to the end of study at 24 weeks
  Inflammatory parameters in blood: Interleukin 6 (pg/ml)
Inflamatory parameters | From enrollment to the end of study at 24 weeks
  Inflammatory parameters in stool: fecal calprotectin (µg/g)
Clinical parameters | From enrollment to the end of study at 24 weeks
  Clinical parameters: gastrointestinal symptoms (abdominal pain: YES/NO; rectal tenesmus: YES/NO; defecatory urge: YES/NO)
Clinical parameters | From enrollment to the end of study at 24 weeks
  Clinical parameters: number and consistency of stools
Clinical parameters | From enrollment to the end of study at 24 weeks
  Clinical parameters: fever (YES/NO), extraintestinal manifestations (YES/NO)
Sarcopenia | From enrollment to the end of study at 24 weeks
  Functional tests (SPPB, measure in seconds)
Sarcopenia | From enrollment to the end of study at 24 weeks
  Dynamometry (kg).
Quality of live and disease remission | From enrollment to the end of study at 24 weeks
  To determine the rate of improvement in the quality of life of patients with using the CVEII9 quality of life.
Quality of live and disease remission | From enrollment to the end of study at 24 weeks
  To determine the rate of the disease remission by evaluating the Crohn's Disease Activity Index (Harvey-Bradshaw Index).
Intestinal microbiota | From enrollment to the end of study at 24 weeks
  To analyze the modifications in the intestinal microbiota resulting from the im-plementation of the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Ramos Molina, Investigator of IMIB, Study Director — Instituto Murciano de Investigación Biosanitaria (IMIB); Antonio J. Ruiz Alcaraz, Investigator of IMIB, Study Director — Instituto Murciano de Investigación Biosanitaria
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided